CLINICAL TRIAL: NCT03943043
Title: A Multicenter, Phase I-II Trial of Gemcitabine Plus Oxaliplatin and Nab-paclitaxel in Subjects With Advanced (Unresectable or Metastatic) Biliary Tract Cancer
Brief Title: Gemcitabine + Oxaliplatin +Nab-paclitaxel in Subjects With Advanced Biliary Tract Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC-2016-001; 2016-004118-84 (EudraCT Number)
Record Dates: First submitted 2018-04-09; First posted 2019-05-09 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — 130-nm albumin-bound paclitaxel; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- gemcitabine oxaliplatin nab-paclitaxel (Experimental): combination at different dose of gemcitabine, oxaliplatin and nab-paclitaxel
  Interventions: Drug: nab-paclitaxel

INTERVENTIONS:
Drug: nab-paclitaxel — Phase I dosing regimens:
  The dose of treatment will be assigned at the time of enrolment in one of these 3 subsequent dose-levels:
  - 1° level: gemcitabine 800 mg/m2 + oxaliplatin 80 mg/m2 + nab-paclitaxel 80 mg/m2 0° level: gemcitabine 1000 mg/m2 + oxaliplatin 80 mg/m2 + nab-paclitaxel 100 mg/m2
  1. level: gemcitabine 1000 mg/m2 + oxaliplatin 80 mg/m2 + nab-paclitaxel 125 mg/m2
  2. level: gemcitabine 1000 mg/m2 + oxaliplatin 80 mg/m2 + nab-paclitaxel 150 mg/m2 each administered on day 1, every 14 day
  Phase II:
  Gemcitabine plus oxaliplatin plus nab-paclitaxel according to RP2D.
  Other Names: Gemcitabine; Oxaliplatin

SUMMARY:
The objective of the study is to determine a new combination of drug that improves the outcome in patients with advanced (unresectable or metastatic) BTC. The primary objective of the phase I part of the study is to determine the maximum tolerated dose (MTD) of the combination gemcitabine plus oxaliplatin plus nab-paclitaxel, established in the first cycle of therapy, in order to determine the recommended phase II dose (RP2D).

The primary objective of the phase II is to determine activity of GEMOX plus nab-paclitaxel. The secondary objectives of the study consist in to better define the safety profile and the outcome of the study treated population.

DETAILED DESCRIPTION:
Systemic chemotherapy is increasingly being applied in cases of biliary tract cancers. A benefit for chemotherapy over best supportive care alone was suggested in a trial that randomly assigned 90 patients with advanced pancreatic or biliary cancer (37 with bile duct cancer) to fluorouracil (FU)-based systemic chemotherapy or best supportive care alone (median survival 6 versus 2.5 months, respectively) (1).

The literature regarding treatment results with specific regimens is limited because most series are small, and many reports consist of a mix of bile duct cancers, gallbladder cancer, ampullary cancer, and either pancreatic or hepatocellular cancers. Although they arise in similar locations, these cancers all have a unique natural history and response to chemotherapy. In general, no single drug or combination has consistently increased median survival beyond the expected six to eight months.

ELIGIBILITY:
Inclusion Criteria:

* Written, signed informed consent
* Male or female aged 18 years or older
* Histologically or citologically-confirmed advanced (unresectable or metastatic) BTC (gallbladder cancer, cancer of the extrahepatic bile duct, intrahepatic cholangiocarcinoma and ampullary carcinoma)
* Measurable or evaluable but non-measurable disease according to RECIST v. 1.1
* Chemotherapy-naïve (prior chemotherapy in the adjuvant setting completed more than 6 months before the trial entry is accepted)
* Adequate bone marrow, liver, and renal function
* ECOG PS 0-1
* Life expectancy of at least 12 weeks
* Negative serum pregnancy test for women of childbearing potential;
* Adoption of adequate contraceptive methods when applicable Women of child-bearing potential must use the following adequate contraceptive methods during all the study and for 1 month after completion of study treatment: abstinence, tubal ligation, oral contraception or transdermal contraceptives, copper intrauterine device, vasectomy of the partner. For male patients with female partners of childbearing potential, agreement to use a barrier method of contraception from the first dose of treatment and for 6 months after completion of study treatment.
* Male patients mustn't donate sperm during the treatment with nab-paclitexel and for 6 months after completion of study treatment.
* Agreement not to donate blood during the study.

Exclusion Criteria:

* Peripheral neuropathy of grade 2 or greater by Common Terminology Criteria for Adverse Events (CTCAE) 4.0. In CTCAE version 4.0 grade 2 sensory neuropathy is defined as moderate symptoms; limiting instrumental activities of daily living (ADLs)
* Previous systemic treatment for advanced disease
* Known symptomatic brain metastases or carcinomatous meningitis
* Severe or uncontrolled systemic disease and/or active or uncontrolled infection
* Women who are currently pregnant or breast feeding
* Previous or current malignancies of other histologies within the last 3 years, with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin
* Known hypersensitivity to nab-paclitaxel, gemcitabine, oxaliplatin or any of the excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2017-07-21 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose | 4 weeks
  Determination of the maximum tolerated dose for phase I

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 16 weeks
  The secondary objectives of the study consist in to better define the safety profile as assessed by CTCAE V4.0
Number of responder (in term of CR, PR, SD) to GEMOX plus nab-paclitaxel as assessed by RECIST 1.1 | Maximum of 24 weeks
  Determination of activity of GEMOX plus nab-paclitaxel as assessed by RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pressiani T, Balsano R, Giordano L, Milella M, Bergamo F, Bozzarelli S, Noventa S, Ferrrari D, Scartozzi M, Parra HS, Auriemma A, Solda C, Zaniboni A, Zecchetto C, Rizzato MD, Rimassa L, Santoro A. Multicenter phase I/II trial of gemcitabine, oxaliplatin and nab-paclitaxel as first-line treatment for patients with advanced biliary tract cancer. Eur J Cancer. 2024 Aug;207:114196. doi: 10.1016/j.ejca.2024.114196. Epub 2024 Jun 29. PMID 38954899